CLINICAL TRIAL: NCT00098566
Title: A Long-Term Follow-Up Study Evaluating the Efficacy and Delayed Toxicities of Radioiodinated Tositumomab (Anti-CD20 Antibody) Followed by Autologous Transplantation for Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Long-Term Effects of Iodine I Tositumomab and Autologous Bone Marrow or Stem Cell Transplantation in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Press, Oliver MD, Fred Hutchinson Cancer Research Center
Other Study IDs: 1734.00; FHCRC-1734.00; CDR0000398806 (Registry Identifier: PDQ)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Lymphoma; Quality of Life
Keywords: quality of life; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent small lymphocytic lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; Waldenstrom macroglobulinemia; recurrent adult grade III lymphomatoid granulomatosis; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
RATIONALE: Studying the long-term effects of cancer treatment in cancer survivors may help improve the ability to plan effective treatment and follow-up care.

PURPOSE: This phase II trial is studying the long-term effects of iodine I 131 tositumomab and autologous bone marrow or stem cell transplantation in patients with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free survival and overall survival of patients with relapsed or refractory B-cell non-Hodgkin's lymphoma previously treated with iodine I^131 tositumomab followed by autologous bone marrow or stem cell transplantation on FHCRC protocols 296, 521, 792, or 915.
* Determine the long-term toxic effects of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a long-term, follow-up study.

Patients undergo testing for human anti-mouse antibody at 1, 3 and 12 months. Patients undergo physical examinations, blood tests, and immune system assessments every 3 months for 1 year and then annually thereafter. Thyroid, pulmonary, and cardiac function are assessed at 1 year and then annually as needed. Patients also undergo CT scans and bone marrow biopsy (if clinically indicated) annually for up to 10 years.

Quality of life is assessed annually.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell non-Hodgkin's lymphoma

  * Relapsed or refractory disease
* Previously treated with myeloablative doses of iodine I^131 tositumomab and autologous bone marrow or stem cell transplantation on 1 of the following phase I or II protocols:

  * FHCRC-296
  * FHCRC-521
  * FHCRC-792
  * FHCRC-915

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated with myeloablative doses of iodine I^131 tositumomab and autologous bone marrow or stem cell transplantation on 1 of the following phase I or II protocols:
  * FHCRC-296
  * FHCRC-521
  * FHCRC-792
  * FHCRC-915
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2002-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Progression-free and overall survival of patients on phase I and II trials by Kaplan Meier survival analyses annually | Annual throughout survival
Toxicity of patients on phase I and II trials by NCI CTC scale annually | Annual throughout survival

CONTACTS AND LOCATIONS:
Overall Officials: Oliver W. Press, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States